CLINICAL TRIAL: NCT02067338
Title: The Effect of Epidural Low-dose Morphine-soaked Microfibrillar Collagen Sponge in Postoperative Pain Control After Posterior Lumbar Spinal Surgery: a Randomized, Double-blind, Placebo-controlled
Brief Title: Epidural Low Dose Morphine in Postoperative Pain After Posterior Lumbar Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SI 387/2012
Record Dates: First submitted 2014-02-09; First posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Morphine
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal saline (Placebo Comparator): During posterior lumbar spinal surgery,one group of patient received normal saline soaked collagen sponge.
  Interventions: Drug: normal saline
- 1 mg morphine soak in epidural oxidized cellulose (Active Comparator): During posterior lumbar spinal surgery ,Another group of patients received 1 mg morphine-soaked in epidural oxidized cellulose.
  Interventions: Drug: 1 mg morphine soak in epidural oxidized cellulose

INTERVENTIONS:
Drug: 1 mg morphine soak in epidural oxidized cellulose — During posterior lumbar spinal surgery , patients received 1 mg morphine-soaked in epidural oxidized cellulose.
  Arms: 1 mg morphine soak in epidural oxidized cellulose
Drug: normal saline — During posterior lumbar spinal surgery , patients received NSS -soaked in epidural oxidized cellulose.
  Arms: normal saline

SUMMARY:
The effect of epidural low-dose morphine-soaked microfibrillar collagen sponge in postoperative pain control after posterior lumbar spinal surgery: a randomized, double-blind, placebo-controlled study

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Yrs
* Good orientation and communication

Exclusion Criteria:

* opioids or sulfonamides allergy
* Contraindication for use
* Epidural morphine
* Selective COX 2 inhibitor
* Patient-controlled analgesia (PCA)
* ASA class > 3
* BMI ≥ 35 kg/sq.m.
* Preoperative use of opioids within 6 Wks
* Intraoperative bleeding > 1000ml

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
VAS measurement was recorded at twenty-four hour after posterior lumbar spinal surgery then compare VAS between low-dose 1 mg morphine-soaked microfibrillar collagen sponge method with normal saline soked | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj hospital, Bangkoknoi, Bangkok, Thailand